CLINICAL TRIAL: NCT02116127
Title: Transcranial Direct Current Stimulation (tDCS) for Depression in Pregnancy: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NI14-020
Record Dates: First submitted 2014-04-02; First posted 2014-04-16 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Depression; Pregnancy
Keywords: Depression; Pregnancy; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): The intervention is active 2mA transcranial direct current stimulation (tDCS). Direct current will be transferred with a pair of saline soaked sponge electrodes (contact area 5 x 7cm), and delivered for 30 minutes. The electrodes will be placed over F3 and F4 according to the 10-20 international system for EEG placement.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): The sham intervention is transcranial direct current stimulation (tDCS). 2mA of direct current will be transferred with a pair of saline soaked sponge electrodes (contact area 5 x 7cm), and the current will be turned off after 54 seconds.The electrodes will be placed over F3 and F4 according to the 10-20 international system for EEG placement.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — The intervention is active 2mA transcranial direct current stimulation (tDCS). Direct current will be transferred with a pair of saline soaked sponge electrodes (contact area 5 x 7cm), and delivered for 30 minutes. The electrodes will be placed over F3 and F4 according to the 10-20 international system for EEG placement.
  Arms: Active tDCS
Device: Sham tDCS — The sham intervention is transcranial direct current stimulation (tDCS). 2mA of direct current will be transferred with a pair of saline soaked sponge electrodes (contact area 5 x 7cm), and the current will be turned off after 54 seconds.The electrodes will be placed over F3 and F4 according to the 10-20 international system for EEG placement.
  Arms: Sham tDCS

SUMMARY:
The purpose of this pilot study is to examine the feasibility of conducting a multi-site double-blind randomized controlled trial whose aim will be to evaluate the effectiveness of transcranial direct current stimulation (tDCS) for treatment in pregnant women with moderate to severe major depression.

DETAILED DESCRIPTION:
Major depression is a serious condition that affects up to 10% of pregnant women, and has serious impact on the developing fetus. However current treatments are less than ideal for women with moderate to severe depression. Psychotherapy alone is either ineffective, or takes months to improve symptoms, leaving the fetus susceptible to depression during that time. Antidepressant medication is effective, but there are high refusal rates of standard pharmacological treatment because of fears about medication exposure. The highly negative impacts of depression in pregnancy on the developing fetus and child illustrate the need for evaluation of timely and innovative treatments.

Transcranial direct current stimulation (tDCS) is a non-drug treatment for depression where the dorsolateral prefrontal cortex, a part of the brain that functions abnormally when an individual is depressed, can be directly stimulated without impacting any other parts of the body or brain. As such, it is an ideal treatment for pregnant women who do not want to expose their fetus to the impact of medication treatment for depression. It has been shown to be effective in depression among non-pregnant adults and improvement is seen rapidly with a 3-week treatment course, almost 3 times faster than standard psychological treatment. There are no known serious adverse effects and no theoretical risk to a fetus.

This research study will measure the feasibility, acceptability and compliance of the tDCS as a treatment option for depression in pregnancy. In addition, the study will investigate the effect of tDCS on reducing depressive symptoms immediately post-treatment among women who have moderate to severe depression in pregnancy.

In this multi-centre, pilot randomized controlled trial, adult women with moderate to severe depression in pregnancy will be recruited from one hospital obstetrical group and two specialty perinatal mental health clinics over the course of 1 year. Women will have been offered to start or continue SSRI (Selective Serotonin Reuptake Inhibitors) or SNRI (Selective Serotonin-Norepinephrine Reuptake Inhibitors)medication but declined use. All participants will continue to receive clinical care from their respective clinical programs during the trial. Although this care may include psychotherapeutic intervention that is initiated prior to completion of the active tDCS treatment phase (if clinic psychotherapy waitlist is short), we would not expect to see improvement within the first 3 weeks of psychotherapeutic treatment. As such, this is an ideal opportunity to evaluate the efficacy of a new treatment, without depriving women of non-pharmacological standard care.

Following informed consent procedures, participants will be randomized to tDCS or a sham-control condition (1:1) with on-site treatments 5 days per week over 3 weeks in 30 minute sessions. The intervention is active 2mA transcranial direct current stimulation (tDCS). Direct current will be transferred with a pair of saline soaked sponge electrodes (contact area 5 x 7cm), and delivered by a specially developed, battery driven constant current stimulator. The electrodes will be placed over F3 and F4 according to the international system for EEG (Electroencephalogram) placement. Sham stimulation will be administered using the same stimulation parameters and at the site of active treatment, but the current will be turned off after 30 seconds.

Women will be interviewed at baseline and then followed during treatment, every four weeks until delivery, and at four and twelve weeks postpartum to allow for measurement of depressive symptoms, pregnancy, delivery, neonatal and infant outcomes. Although baseline and treatment interviews will be conducted in person, post-treatment and post-delivery interviews will be offered in person or over the telephone, according to participant preference.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged > 18 years
2. >12 weeks gestation at enrollment
3. 32 or fewer weeks gestation at first treatment visit (to increase likelihood of all treatment occurring during pregnancy)
4. Diagnosis of Major Depressive Disorder and in a Moderate-severe major depressive episode without psychotic features (as confirmed by the Mini-International Neuropsychiatric Interview, MINI ).
5. Safe for outpatient psychiatric treatment (as assessed by Study PI).
6. Offered, but declined to use an anti-depressant medication
7. Capable to consent to treatment
8. Able to understand study explanations and have questionnaires administered in English

Exclusion Criteria:

1. DSM-V history of alcohol and/or substance use or dependence in the previous 6 months
2. Concomitant major and unstable medical or neurologic illness or history of seizure
3. Currently taking carbamazepine (which may interfere with the effects of anodal tDCS),
4. Major complications and/or a known fetal anomaly in the current pregnancy as determined by the investigator team
5. Planning to leave Toronto prior to delivery in the current pregnancy.
6. Metal implant(s) in cranium
7. Electrical implant(s) in body
8. Currently taking benzodiazepines daily (Intermittent PRN use of low-dose Lorazepam allowed)
9. Non-intact skin on scalp areas where stimulation electrodes will be placed
10. History of very preterm delivery in previous pregnancy (< 32 weeks gestation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited over 1 year | Up to one year from when the study starts enrolling participants
  Feasibility

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | End of week 1
  Efficacy - Depression Symptom Measurement
Edinburgh Postnatal Depression Scale | End of Week 1
  Efficacy - Depression Symptom Measurement
Pregnancy Experience Scale | End of Week 1
  Efficacy - Secondary Symptom Measurement
State-Trait Anxiety Inventory | End of week 1
  Efficacy - Secondary Symptom Measurement
Itemized neonatal health outcomes questionnaire | 4 weeks postpartum
  Neonatal outcome (safety)
Itemized neonatal health outcomes questionnaire | 12 weeks postpartum
  Neonatal Outcome (safety)
Bates Infant Characteristics Questionnaire | 12 weeks postpartum
  Infant outcome (temperament)
Ages and Stages Questionnaire | 12 weeks postpartum
  Infant outcome (development)
Toronto Side Effects Scale | End of Week 1
  Acceptability - side effects
Toronto Side Effects Scale | End of week 2
  Acceptability - side effects
Toronto Side Effects Scale | End of intervention phase (end of week 3)
  Acceptability - side effects
Itemized treatment acceptability questionnaire | End of intervention phase (end of week 3)
  Acceptability - barriers and facilitators of attending appointments
Pregnancy Complications Itemized Questionnaire | End of week 1
Pregnancy Complications Itemized Questionnaire | End of week 2
Pregnancy Complications Itemized Questionnaire | End of intervention phase (end of week 3)
Pregnancy Complications Itemized Questionnaire | Every 4 weeks until delivery of baby (up to 26 weeks from initial randomization)
Pregnancy Complications Itemized Questionnaire | 4 weeks postpartum
Rate of follow-up data collection | 12 weeks postpartum
Completion of all 15 treatment sessions | End of intervention phase (end of week 3)
Treatment allocation questionnaire | End of week 1
Treatment allocation questionnaire | End of intervention phase (end of week 3)
Montgomery Asberg Depression Rating Scale | End of week 2
  Efficacy - Depression Symptom Measurement
Edinburgh Postnatal Depression Scale | End of Week 2
  Efficacy - Depression Symptom Measurement
Montgomery Asberg Depression Rating Scale | End of intervention phase (End of week 3)
  Efficacy - Depression Symptom Measurement
Montgomery Asberg Depression Rating Scale | Every 4 weeks until delivery (i.e. up to 26 weeks from initial randomization)
  Efficacy - Depression Symptom Measurement
Montgomery Asberg Depression Rating Scale | 4 weeks postpartum
  Efficacy - Depression Symptom Measurement
Montgomery Asberg Depression Rating Scale | 12 weeks postpartum
  Efficacy - Depression Symptom Measurement
Edinburgh Postnatal Depression Scale | End of intervention phase (Week 3)
  Efficacy - Depression Symptom Measurement
Edinburgh Postnatal Depression Scale | Every 4 weeks until delivery (i.e. up to 26 weeks from initial randomization)
  Efficacy - Depression Symptom Measurement
Edinburgh Postnatal Depression Scale | 4 weeks postpartum
  Efficacy - Depression Symptom Measurement
Edinburgh Postnatal Depression Scale | 12 weeks postpartum
  Efficacy - Depression Symptom Measurement
Pregnancy Experience Scale | End of Week 2
  Efficacy - Secondary Symptom Measurement
Pregnancy Experience Scale | End of intervention phase (Week 3)
  Efficacy - Secondary Symptom Measurement
Pregnancy Experience Scale | Every 4 weeks until delivery (i.e. up to 26 weeks from initial randomization)
  Efficacy - Secondary Symptom Measurement
State-Trait Anxiety Inventory | End of week 2
  Efficacy - Secondary Symptom Measurement
State-Trait Anxiety Inventory | End of intervention phase (end of week 3)
  Efficacy - Secondary Symptom Measurement
State-Trait Anxiety Inventory | Every 4 weeks until delivery (i.e. up to 26 weeks from initial randomization)
  Efficacy - Secondary Symptom Measurement
State-Trait Anxiety Inventory | 4 weeks postpartum
  Efficacy - Secondary Symptom Measurement
State-Trait Anxiety Inventory | 12 weeks postpartum
  Efficacy - Secondary Symptom Measurement

CONTACTS AND LOCATIONS:
Overall Officials: Simone N Vigod, MD, MSc, Principal Investigator — Women's College Hospital; Daniel M Blumberger, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

REFERENCES:
- [Background] Bates JE, Freeland CA, Lounsbury ML. Measurement of infant difficultness. Child Dev. 1979 Sep;50(3):794-803. PMID 498854
- [Background] Steer RA, Scholl TO, Hediger ML, Fischer RL. Self-reported depression and negative pregnancy outcomes. J Clin Epidemiol. 1992 Oct;45(10):1093-9. doi: 10.1016/0895-4356(92)90149-h. PMID 1474405
- [Background] Murray L. The impact of postnatal depression on infant development. J Child Psychol Psychiatry. 1992 Mar;33(3):543-61. doi: 10.1111/j.1469-7610.1992.tb00890.x. PMID 1577898
- [Background] Zuckerman B, Bauchner H, Parker S, Cabral H. Maternal depressive symptoms during pregnancy, and newborn irritability. J Dev Behav Pediatr. 1990 Aug;11(4):190-4. PMID 2212032
- [Background] Williams JB. A structured interview guide for the Hamilton Depression Rating Scale. Arch Gen Psychiatry. 1988 Aug;45(8):742-7. doi: 10.1001/archpsyc.1988.01800320058007. PMID 3395203
- [Background] Sandman CA, Wadhwa PD, Dunkel-Schetter C, Chicz-DeMet A, Belman J, Porto M, Murata Y, Garite TJ, Crinella FM. Psychobiological influences of stress and HPA regulation on the human fetus and infant birth outcomes. Ann N Y Acad Sci. 1994 Oct 31;739:198-210. doi: 10.1111/j.1749-6632.1994.tb19822.x. No abstract available. PMID 7832474
- [Background] Pastuszak A, Schick-Boschetto B, Zuber C, Feldkamp M, Pinelli M, Sihn S, Donnenfeld A, McCormack M, Leen-Mitchell M, Woodland C, et al. Pregnancy outcome following first-trimester exposure to fluoxetine (Prozac). JAMA. 1993 May 5;269(17):2246-8. PMID 8474204
- [Background] Orr ST, Miller CA. Maternal depressive symptoms and the risk of poor pregnancy outcome. Review of the literature and preliminary findings. Epidemiol Rev. 1995;17(1):165-71. doi: 10.1093/oxfordjournals.epirev.a036172. No abstract available. PMID 8521934
- [Background] Chambers CD, Johnson KA, Dick LM, Felix RJ, Jones KL. Birth outcomes in pregnant women taking fluoxetine. N Engl J Med. 1996 Oct 3;335(14):1010-5. doi: 10.1056/NEJM199610033351402. PMID 8793924
- [Background] Kulin NA, Pastuszak A, Sage SR, Schick-Boschetto B, Spivey G, Feldkamp M, Ormond K, Matsui D, Stein-Schechman AK, Cook L, Brochu J, Rieder M, Koren G. Pregnancy outcome following maternal use of the new selective serotonin reuptake inhibitors: a prospective controlled multicenter study. JAMA. 1998 Feb 25;279(8):609-10. doi: 10.1001/jama.279.8.609. PMID 9486756
- [Background] Beck CT. The effects of postpartum depression on child development: a meta-analysis. Arch Psychiatr Nurs. 1998 Feb;12(1):12-20. doi: 10.1016/s0883-9417(98)80004-6. PMID 9489170
- [Background] Sinclair D, Murray L. Effects of postnatal depression on children's adjustment to school. Teacher's reports. Br J Psychiatry. 1998 Jan;172:58-63. doi: 10.1192/bjp.172.1.58. PMID 9534834
- [Background] Weinberg MK, Tronick EZ. The impact of maternal psychiatric illness on infant development. J Clin Psychiatry. 1998;59 Suppl 2:53-61. PMID 9559760
- [Background] Judd LL, Akiskal HS, Maser JD, Zeller PJ, Endicott J, Coryell W, Paulus MP, Kunovac JL, Leon AC, Mueller TI, Rice JA, Keller MB. A prospective 12-year study of subsyndromal and syndromal depressive symptoms in unipolar major depressive disorders. Arch Gen Psychiatry. 1998 Aug;55(8):694-700. doi: 10.1001/archpsyc.55.8.694. PMID 9707379
- [Background] Teixeira JM, Fisk NM, Glover V. Association between maternal anxiety in pregnancy and increased uterine artery resistance index: cohort based study. BMJ. 1999 Jan 16;318(7177):153-7. doi: 10.1136/bmj.318.7177.153. PMID 9888905
- [Background] Ericson A, Kallen B, Wiholm B. Delivery outcome after the use of antidepressants in early pregnancy. Eur J Clin Pharmacol. 1999 Sep;55(7):503-8. doi: 10.1007/s002280050664. PMID 10501819
- [Background] Martins C, Gaffan EA. Effects of early maternal depression on patterns of infant-mother attachment: a meta-analytic investigation. J Child Psychol Psychiatry. 2000 Sep;41(6):737-46. PMID 11039686
- [Background] Cohen LS, Heller VL, Bailey JW, Grush L, Ablon JS, Bouffard SM. Birth outcomes following prenatal exposure to fluoxetine. Biol Psychiatry. 2000 Nov 15;48(10):996-1000. doi: 10.1016/s0006-3223(00)00877-5. PMID 11082474
- [Background] Michaud CM, Murray CJ, Bloom BR. Burden of disease--implications for future research. JAMA. 2001 Feb 7;285(5):535-9. doi: 10.1001/jama.285.5.535. PMID 11176854
- [Background] Speer AM, Kimbrell TA, Wassermann EM, D Repella J, Willis MW, Herscovitch P, Post RM. Opposite effects of high and low frequency rTMS on regional brain activity in depressed patients. Biol Psychiatry. 2000 Dec 15;48(12):1133-41. doi: 10.1016/s0006-3223(00)01065-9. PMID 11137053
- [Background] Uno H, Lohmiller L, Thieme C, Kemnitz JW, Engle MJ, Roecker EB, Farrell PM. Brain damage induced by prenatal exposure to dexamethasone in fetal rhesus macaques. I. Hippocampus. Brain Res Dev Brain Res. 1990 May 1;53(2):157-67. doi: 10.1016/0165-3806(90)90002-g. PMID 2357788
- [Background] Stiskal JA, Kulin N, Koren G, Ho T, Ito S. Neonatal paroxetine withdrawal syndrome. Arch Dis Child Fetal Neonatal Ed. 2001 Mar;84(2):F134-5. doi: 10.1136/fn.84.2.f134. PMID 11207233
- [Background] Nordeng H, Lindemann R, Perminov KV, Reikvam A. Neonatal withdrawal syndrome after in utero exposure to selective serotonin reuptake inhibitors. Acta Paediatr. 2001 Mar;90(3):288-91. PMID 11332169
- [Background] Herwig U, Padberg F, Unger J, Spitzer M, Schonfeldt-Lecuona C. Transcranial magnetic stimulation in therapy studies: examination of the reliability of "standard" coil positioning by neuronavigation. Biol Psychiatry. 2001 Jul 1;50(1):58-61. doi: 10.1016/s0006-3223(01)01153-2. PMID 11457424
- [Background] Hasey G. Transcranial magnetic stimulation in the treatment of mood disorder: a review and comparison with electroconvulsive therapy. Can J Psychiatry. 2001 Oct;46(8):720-7. doi: 10.1177/070674370104600804. PMID 11692974
- [Background] Oberlander TF, Eckstein Grunau R, Fitzgerald C, Ellwood AL, Misri S, Rurak D, Riggs KW. Prolonged prenatal psychotropic medication exposure alters neonatal acute pain response. Pediatr Res. 2002 Apr;51(4):443-53. doi: 10.1203/00006450-200204000-00008. PMID 11919328
- [Background] Kelly RH, Russo J, Holt VL, Danielsen BH, Zatzick DF, Walker E, Katon W. Psychiatric and substance use disorders as risk factors for low birth weight and preterm delivery. Obstet Gynecol. 2002 Aug;100(2):297-304. doi: 10.1016/s0029-7844(02)02014-8. PMID 12151153
- [Background] Sharma V. Pharmacotherapy of postpartum depression. Expert Opin Pharmacother. 2002 Oct;3(10):1421-31. doi: 10.1517/14656566.3.10.1421. PMID 12387688
- [Background] Nulman I, Rovet J, Stewart DE, Wolpin J, Pace-Asciak P, Shuhaiber S, Koren G. Child development following exposure to tricyclic antidepressants or fluoxetine throughout fetal life: a prospective, controlled study. Am J Psychiatry. 2002 Nov;159(11):1889-95. doi: 10.1176/appi.ajp.159.11.1889. PMID 12411224
- [Background] Costei AM, Kozer E, Ho T, Ito S, Koren G. Perinatal outcome following third trimester exposure to paroxetine. Arch Pediatr Adolesc Med. 2002 Nov;156(11):1129-32. doi: 10.1001/archpedi.156.11.1129. PMID 12413342
- [Background] Simon GE, Cunningham ML, Davis RL. Outcomes of prenatal antidepressant exposure. Am J Psychiatry. 2002 Dec;159(12):2055-61. doi: 10.1176/appi.ajp.159.12.2055. PMID 12450956
- [Background] Nitsche MA. Transcranial direct current stimulation: a new treatment for depression? Bipolar Disord. 2002;4 Suppl 1:98-9. doi: 10.1034/j.1399-5618.4.s1.43.x. No abstract available. PMID 12479691
- [Background] Hammen C, Brennan PA. Severity, chronicity, and timing of maternal depression and risk for adolescent offspring diagnoses in a community sample. Arch Gen Psychiatry. 2003 Mar;60(3):253-8. doi: 10.1001/archpsyc.60.3.253. PMID 12622658
- [Background] Dennis CL. The effect of peer support on postpartum depression: a pilot randomized controlled trial. Can J Psychiatry. 2003 Mar;48(2):115-24. doi: 10.1177/070674370304800209. PMID 12655910
- [Background] Casper RC, Fleisher BE, Lee-Ancajas JC, Gilles A, Gaylor E, DeBattista A, Hoyme HE. Follow-up of children of depressed mothers exposed or not exposed to antidepressant drugs during pregnancy. J Pediatr. 2003 Apr;142(4):402-8. doi: 10.1067/mpd.2003.139. PMID 12712058
- [Background] Laine K, Heikkinen T, Ekblad U, Kero P. Effects of exposure to selective serotonin reuptake inhibitors during pregnancy on serotonergic symptoms in newborns and cord blood monoamine and prolactin concentrations. Arch Gen Psychiatry. 2003 Jul;60(7):720-6. doi: 10.1001/archpsyc.60.7.720. PMID 12860776
- [Background] Fitzgerald PB, Brown TL, Marston NA, Daskalakis ZJ, De Castella A, Kulkarni J. Transcranial magnetic stimulation in the treatment of depression: a double-blind, placebo-controlled trial. Arch Gen Psychiatry. 2003 Oct;60(10):1002-8. doi: 10.1001/archpsyc.60.9.1002. PMID 14557145
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Gjerdingen D. The effectiveness of various postpartum depression treatments and the impact of antidepressant drugs on nursing infants. J Am Board Fam Pract. 2003 Sep-Oct;16(5):372-82. doi: 10.3122/jabfm.16.5.372. PMID 14645327
- [Background] Lang N, Nitsche MA, Paulus W, Rothwell JC, Lemon RN. Effects of transcranial direct current stimulation over the human motor cortex on corticospinal and transcallosal excitability. Exp Brain Res. 2004 Jun;156(4):439-43. doi: 10.1007/s00221-003-1800-2. Epub 2004 Jan 24. PMID 14745467
- [Background] Bennett HA, Einarson A, Taddio A, Koren G, Einarson TR. Prevalence of depression during pregnancy: systematic review. Obstet Gynecol. 2004 Apr;103(4):698-709. doi: 10.1097/01.AOG.0000116689.75396.5f. PMID 15051562
- [Background] Dennis CL. Preventing postpartum depression part I: a review of biological interventions. Can J Psychiatry. 2004 Jul;49(7):467-75. doi: 10.1177/070674370404900708. PMID 15362251
- [Background] Dennis CL, Stewart DE. Treatment of postpartum depression, part 1: a critical review of biological interventions. J Clin Psychiatry. 2004 Sep;65(9):1242-51. doi: 10.4088/jcp.v65n0914. PMID 15367053
- [Background] Dennis CL. Treatment of postpartum depression, part 2: a critical review of nonbiological interventions. J Clin Psychiatry. 2004 Sep;65(9):1252-65. doi: 10.4088/jcp.v65n0915. PMID 15367054
- [Background] Dennis CL. Preventing postpartum depression part II: A critical review of nonbiological interventions. Can J Psychiatry. 2004 Aug;49(8):526-38. doi: 10.1177/070674370404900804. PMID 15453102
- [Background] Fitzgerald PB, Brown TL, Marston NA, Daskalakis ZJ, de Castella A, Bradshaw JL, Kulkarni J. Motor cortical excitability and clinical response to rTMS in depression. J Affect Disord. 2004 Oct 1;82(1):71-6. doi: 10.1016/j.jad.2003.09.014. PMID 15465578
- [Background] DiPietro JA, Ghera MM, Costigan K, Hawkins M. Measuring the ups and downs of pregnancy stress. J Psychosom Obstet Gynaecol. 2004 Sep-Dec;25(3-4):189-201. doi: 10.1080/01674820400017830. PMID 15715018
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Ardolino G, Bossi B, Barbieri S, Priori A. Non-synaptic mechanisms underlie the after-effects of cathodal transcutaneous direct current stimulation of the human brain. J Physiol. 2005 Oct 15;568(Pt 2):653-63. doi: 10.1113/jphysiol.2005.088310. Epub 2005 Jul 21. PMID 16037080
- [Background] Fregni F, Boggio PS, Mansur CG, Wagner T, Ferreira MJ, Lima MC, Rigonatti SP, Marcolin MA, Freedman SD, Nitsche MA, Pascual-Leone A. Transcranial direct current stimulation of the unaffected hemisphere in stroke patients. Neuroreport. 2005 Sep 28;16(14):1551-5. doi: 10.1097/01.wnr.0000177010.44602.5e. PMID 16148743
- [Background] Pilowsky DJ, Wickramaratne PJ, Rush AJ, Hughes CW, Garber J, Malloy E, King CA, Cerda G, Sood AB, Alpert JE, Wisniewski SR, Trivedi MH, Talati A, Carlson MM, Liu HH, Fava M, Weissman MM. Children of currently depressed mothers: a STAR*D ancillary study. J Clin Psychiatry. 2006 Jan;67(1):126-36. doi: 10.4088/jcp.v67n0119. PMID 16426099
- [Background] Cohen LS, Altshuler LL, Harlow BL, Nonacs R, Newport DJ, Viguera AC, Suri R, Burt VK, Hendrick V, Reminick AM, Loughead A, Vitonis AF, Stowe ZN. Relapse of major depression during pregnancy in women who maintain or discontinue antidepressant treatment. JAMA. 2006 Feb 1;295(5):499-507. doi: 10.1001/jama.295.5.499. PMID 16449615
- [Background] Levinson-Castiel R, Merlob P, Linder N, Sirota L, Klinger G. Neonatal abstinence syndrome after in utero exposure to selective serotonin reuptake inhibitors in term infants. Arch Pediatr Adolesc Med. 2006 Feb;160(2):173-6. doi: 10.1001/archpedi.160.2.173. PMID 16461873
- [Background] Chambers CD, Hernandez-Diaz S, Van Marter LJ, Werler MM, Louik C, Jones KL, Mitchell AA. Selective serotonin-reuptake inhibitors and risk of persistent pulmonary hypertension of the newborn. N Engl J Med. 2006 Feb 9;354(6):579-87. doi: 10.1056/NEJMoa052744. PMID 16467545
- [Background] Fregni F, Boggio PS, Nitsche MA, Marcolin MA, Rigonatti SP, Pascual-Leone A. Treatment of major depression with transcranial direct current stimulation. Bipolar Disord. 2006 Apr;8(2):203-4. doi: 10.1111/j.1399-5618.2006.00291.x. No abstract available. PMID 16542193
- [Background] Weissman MM, Pilowsky DJ, Wickramaratne PJ, Talati A, Wisniewski SR, Fava M, Hughes CW, Garber J, Malloy E, King CA, Cerda G, Sood AB, Alpert JE, Trivedi MH, Rush AJ; STAR*D-Child Team. Remissions in maternal depression and child psychopathology: a STAR*D-child report. JAMA. 2006 Mar 22;295(12):1389-98. doi: 10.1001/jama.295.12.1389. PMID 16551710
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Wen SW, Yang Q, Garner P, Fraser W, Olatunbosun O, Nimrod C, Walker M. Selective serotonin reuptake inhibitors and adverse pregnancy outcomes. Am J Obstet Gynecol. 2006 Apr;194(4):961-6. doi: 10.1016/j.ajog.2006.02.019. PMID 16580283
- [Background] Miranda PC, Lomarev M, Hallett M. Modeling the current distribution during transcranial direct current stimulation. Clin Neurophysiol. 2006 Jul;117(7):1623-9. doi: 10.1016/j.clinph.2006.04.009. Epub 2006 Jun 9. PMID 16762592
- [Background] Boggio PS, Castro LO, Savagim EA, Braite R, Cruz VC, Rocha RR, Rigonatti SP, Silva MT, Fregni F. Enhancement of non-dominant hand motor function by anodal transcranial direct current stimulation. Neurosci Lett. 2006 Aug 14;404(1-2):232-6. doi: 10.1016/j.neulet.2006.05.051. Epub 2006 Jun 30. PMID 16808997
- [Background] Fitzgerald PB, Benitez J, de Castella AR, Brown TL, Daskalakis ZJ, Kulkarni J. Naturalistic study of the use of transcranial magnetic stimulation in the treatment of depressive relapse. Aust N Z J Psychiatry. 2006 Sep;40(9):764-8. doi: 10.1080/j.1440-1614.2006.01881.x. PMID 16911751
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Loo CK, McFarquhar TF, Mitchell PB. A review of the safety of repetitive transcranial magnetic stimulation as a clinical treatment for depression. Int J Neuropsychopharmacol. 2008 Feb;11(1):131-47. doi: 10.1017/S1461145707007717. Epub 2007 Sep 20. PMID 17880752
- [Background] Marcus SM, Flynn HA. Depression, antidepressant medication, and functioning outcomes among pregnant women. Int J Gynaecol Obstet. 2008 Mar;100(3):248-51. doi: 10.1016/j.ijgo.2007.09.016. Epub 2007 Nov 19. PMID 18005968
- [Background] Pilowsky DJ, Wickramaratne P, Talati A, Tang M, Hughes CW, Garber J, Malloy E, King C, Cerda G, Sood AB, Alpert JE, Trivedi MH, Fava M, Rush AJ, Wisniewski S, Weissman MM. Children of depressed mothers 1 year after the initiation of maternal treatment: findings from the STAR*D-Child Study. Am J Psychiatry. 2008 Sep;165(9):1136-47. doi: 10.1176/appi.ajp.2008.07081286. Epub 2008 Jun 16. PMID 18558646
- [Background] Flynn HA, Chermack ST. Prenatal alcohol use: the role of lifetime problems with alcohol, drugs, depression, and violence. J Stud Alcohol Drugs. 2008 Jul;69(4):500-9. doi: 10.15288/jsad.2008.69.500. PMID 18612565
- [Background] Dennis CL, Allen K. Interventions (other than pharmacological, psychosocial or psychological) for treating antenatal depression. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006795. doi: 10.1002/14651858.CD006795.pub2. PMID 18843730
- [Background] Anderson EL, Reti IM. ECT in pregnancy: a review of the literature from 1941 to 2007. Psychosom Med. 2009 Feb;71(2):235-42. doi: 10.1097/PSY.0b013e318190d7ca. Epub 2008 Dec 10. PMID 19073751
- [Background] Fitzgerald PB, Hoy K, McQueen S, Maller JJ, Herring S, Segrave R, Bailey M, Been G, Kulkarni J, Daskalakis ZJ. A randomized trial of rTMS targeted with MRI based neuro-navigation in treatment-resistant depression. Neuropsychopharmacology. 2009 Apr;34(5):1255-62. doi: 10.1038/npp.2008.233. Epub 2009 Jan 14. PMID 19145228
- [Background] Marcus SM. Depression during pregnancy: rates, risks and consequences--Motherisk Update 2008. Can J Clin Pharmacol. 2009 Winter;16(1):e15-22. Epub 2009 Jan 22. PMID 19164843
- [Background] Wisner KL, Sit DK, Hanusa BH, Moses-Kolko EL, Bogen DL, Hunker DF, Perel JM, Jones-Ivy S, Bodnar LM, Singer LT. Major depression and antidepressant treatment: impact on pregnancy and neonatal outcomes. Am J Psychiatry. 2009 May;166(5):557-66. doi: 10.1176/appi.ajp.2008.08081170. Epub 2009 Mar 16. PMID 19289451
- [Background] Gibson J, McKenzie-McHarg K, Shakespeare J, Price J, Gray R. A systematic review of studies validating the Edinburgh Postnatal Depression Scale in antepartum and postpartum women. Acta Psychiatr Scand. 2009 May;119(5):350-64. doi: 10.1111/j.1600-0447.2009.01363.x. Epub 2009 Mar 2. PMID 19298573
- [Background] Nitsche MA, Boggio PS, Fregni F, Pascual-Leone A. Treatment of depression with transcranial direct current stimulation (tDCS): a review. Exp Neurol. 2009 Sep;219(1):14-9. doi: 10.1016/j.expneurol.2009.03.038. Epub 2009 Apr 5. PMID 19348793
- [Background] Merzagora AC, Foffani G, Panyavin I, Mordillo-Mateos L, Aguilar J, Onaral B, Oliviero A. Prefrontal hemodynamic changes produced by anodal direct current stimulation. Neuroimage. 2010 Feb 1;49(3):2304-10. doi: 10.1016/j.neuroimage.2009.10.044. Epub 2009 Oct 21. PMID 19853048
- [Background] Oberlander TF, Gingrich JA, Ansorge MS. Sustained neurobehavioral effects of exposure to SSRI antidepressants during development: molecular to clinical evidence. Clin Pharmacol Ther. 2009 Dec;86(6):672-7. doi: 10.1038/clpt.2009.201. Epub 2009 Nov 4. PMID 19890255
- [Background] Dennis CL. Postpartum depression peer support: maternal perceptions from a randomized controlled trial. Int J Nurs Stud. 2010 May;47(5):560-8. doi: 10.1016/j.ijnurstu.2009.10.015. Epub 2009 Dec 4. PMID 19962699
- [Background] You JJ, Alter DA, Stukel TA, McDonald SD, Laupacis A, Liu Y, Ray JG. Proliferation of prenatal ultrasonography. CMAJ. 2010 Feb 9;182(2):143-51. doi: 10.1503/cmaj.090979. Epub 2010 Jan 4. PMID 20048009
- [Background] Vigod SN, Villegas L, Dennis CL, Ross LE. Prevalence and risk factors for postpartum depression among women with preterm and low-birth-weight infants: a systematic review. BJOG. 2010 Apr;117(5):540-50. doi: 10.1111/j.1471-0528.2009.02493.x. Epub 2010 Jan 29. PMID 20121831
- [Background] Ross LE, McQueen K, Vigod S, Dennis CL. Risk for postpartum depression associated with assisted reproductive technologies and multiple births: a systematic review. Hum Reprod Update. 2011 Jan-Feb;17(1):96-106. doi: 10.1093/humupd/dmq025. Epub 2010 Jul 6. PMID 20605900
- [Background] Ray JG, Schull MJ, Urquia ML, You JJ, Guttmann A, Vermeulen MJ. Major radiodiagnostic imaging in pregnancy and the risk of childhood malignancy: a population-based cohort study in Ontario. PLoS Med. 2010 Sep 7;7(9):e1000337. doi: 10.1371/journal.pmed.1000337. PMID 20838660
- [Background] Brunoni AR, Valiengo L, Baccaro A, Zanao TA, de Oliveira JF, Vieira GP, Bueno VF, Goulart AC, Boggio PS, Lotufo PA, Bensenor IM, Fregni F. Sertraline vs. ELectrical Current Therapy for Treating Depression Clinical Trial--SELECT TDCS: design, rationale and objectives. Contemp Clin Trials. 2011 Jan;32(1):90-8. doi: 10.1016/j.cct.2010.09.007. Epub 2010 Sep 18. PMID 20854930
- [Background] Wickramaratne P, Gameroff MJ, Pilowsky DJ, Hughes CW, Garber J, Malloy E, King C, Cerda G, Sood AB, Alpert JE, Trivedi MH, Fava M, Rush AJ, Wisniewski S, Weissman MM. Children of depressed mothers 1 year after remission of maternal depression: findings from the STAR*D-Child study. Am J Psychiatry. 2011 Jun;168(6):593-602. doi: 10.1176/appi.ajp.2010.10010032. Epub 2011 Mar 15. PMID 21406462
- [Background] Yonkers KA, Vigod S, Ross LE. Diagnosis, pathophysiology, and management of mood disorders in pregnant and postpartum women. Obstet Gynecol. 2011 Apr;117(4):961-977. doi: 10.1097/AOG.0b013e31821187a7. PMID 21422871
- [Background] Rurak D, Lim K, Sanders A, Brain U, Riggs W, Oberlander TF. Third trimester fetal heart rate and Doppler middle cerebral artery blood flow velocity characteristics during prenatal selective serotonin reuptake inhibitor exposure. Pediatr Res. 2011 Jul;70(1):96-101. doi: 10.1203/PDR.0b013e31821ba11a. PMID 21436759
- [Background] Mulder EJ, Ververs FF, de Heus R, Visser GH. Selective serotonin reuptake inhibitors affect neurobehavioral development in the human fetus. Neuropsychopharmacology. 2011 Sep;36(10):1961-71. doi: 10.1038/npp.2011.67. Epub 2011 Apr 27. PMID 21525859
- [Background] Blumberger DM, Mulsant BH, Fitzgerald PB, Rajji TK, Ravindran AV, Young LT, Levinson AJ, Daskalakis ZJ. A randomized double-blind sham-controlled comparison of unilateral and bilateral repetitive transcranial magnetic stimulation for treatment-resistant major depression. World J Biol Psychiatry. 2012 Sep;13(6):423-35. doi: 10.3109/15622975.2011.579163. Epub 2011 Jul 8. PMID 21736507
- [Background] Raimundo RJS, Uribe CE, Brasil-Neto JP. Lack of clinically detectable acute changes on autonomic or thermoregulatory functions in healthy subjects after transcranial direct current stimulation (tDCS). Brain Stimul. 2012 Jul;5(3):196-200. doi: 10.1016/j.brs.2011.03.009. Epub 2011 Apr 27. PMID 22037121
- [Background] Loo CK, Alonzo A, Martin D, Mitchell PB, Galvez V, Sachdev P. Transcranial direct current stimulation for depression: 3-week, randomised, sham-controlled trial. Br J Psychiatry. 2012 Jan;200(1):52-9. doi: 10.1192/bjp.bp.111.097634. PMID 22215866
- [Background] Kalu UG, Sexton CE, Loo CK, Ebmeier KP. Transcranial direct current stimulation in the treatment of major depression: a meta-analysis. Psychol Med. 2012 Sep;42(9):1791-800. doi: 10.1017/S0033291711003059. Epub 2012 Jan 12. PMID 22236735
- [Background] Blumberger DM, Christensen BK, Zipursky RB, Moller B, Chen R, Fitzgerald PB, Daskalakis ZJ. MRI-targeted repetitive transcranial magnetic stimulation of Heschl's gyrus for refractory auditory hallucinations. Brain Stimul. 2012 Oct;5(4):577-85. doi: 10.1016/j.brs.2011.12.002. Epub 2012 Feb 22. PMID 22410480
- [Background] Dennis CL, Ravitz P, Grigoriadis S, Jovellanos M, Hodnett E, Ross L, Zupancic J. The effect of telephone-based interpersonal psychotherapy for the treatment of postpartum depression: study protocol for a randomized controlled trial. Trials. 2012 Apr 19;13:38. doi: 10.1186/1745-6215-13-38. PMID 22515528
- [Background] Brunoni AR, Vanderhasselt MA, Boggio PS, Fregni F, Dantas EM, Mill JG, Lotufo PA, Bensenor IM. Polarity- and valence-dependent effects of prefrontal transcranial direct current stimulation on heart rate variability and salivary cortisol. Psychoneuroendocrinology. 2013 Jan;38(1):58-66. doi: 10.1016/j.psyneuen.2012.04.020. Epub 2012 May 22. PMID 22626867
- [Background] Fitzgerald PB, Grace N, Hoy KE, Bailey M, Daskalakis ZJ. An open label trial of clustered maintenance rTMS for patients with refractory depression. Brain Stimul. 2013 May;6(3):292-7. doi: 10.1016/j.brs.2012.05.003. Epub 2012 Jun 1. PMID 22683273
- [Background] Hanley GE, Oberlander TF. Neurodevelopmental outcomes following prenatal exposure to serotonin reuptake inhibitor antidepressants: a "social teratogen" or moderator of developmental risk? Birth Defects Res A Clin Mol Teratol. 2012 Aug;94(8):651-9. doi: 10.1002/bdra.23032. Epub 2012 Jun 26. PMID 22733632
- [Background] Blumberger DM, Tran LC, Fitzgerald PB, Hoy KE, Daskalakis ZJ. A randomized double-blind sham-controlled study of transcranial direct current stimulation for treatment-resistant major depression. Front Psychiatry. 2012 Aug 17;3:74. doi: 10.3389/fpsyt.2012.00074. eCollection 2012. PMID 22912618
- [Background] Weikum WM, Oberlander TF, Hensch TK, Werker JF. Prenatal exposure to antidepressants and depressed maternal mood alter trajectory of infant speech perception. Proc Natl Acad Sci U S A. 2012 Oct 16;109 Suppl 2(Suppl 2):17221-7. doi: 10.1073/pnas.1121263109. Epub 2012 Oct 8. PMID 23045665
- [Background] Dennis CL, Heaman M, Vigod S. Epidemiology of postpartum depressive symptoms among Canadian women: regional and national results from a cross-sectional survey. Can J Psychiatry. 2012 Sep;57(9):537-46. doi: 10.1177/070674371205700904. PMID 23073031
- [Background] Seitz DP, Vigod SN, Lin E, Gruneir A, Newman A, Anderson G, Rapoport MJ, Rochon P, Blumberger DM, Herrmann N. Characteristics of older adults hospitalized in acute psychiatric units in ontario: a population-based study. Can J Psychiatry. 2012 Sep;57(9):554-63. doi: 10.1177/070674371205700906. PMID 23073033
- [Background] Nulman I, Koren G, Rovet J, Barrera M, Pulver A, Streiner D, Feldman B. Neurodevelopment of children following prenatal exposure to venlafaxine, selective serotonin reuptake inhibitors, or untreated maternal depression. Am J Psychiatry. 2012 Nov;169(11):1165-74. doi: 10.1176/appi.ajp.2012.11111721. PMID 23128923
- [Background] Byatt N, Simas TA, Lundquist RS, Johnson JV, Ziedonis DM. Strategies for improving perinatal depression treatment in North American outpatient obstetric settings. J Psychosom Obstet Gynaecol. 2012 Dec;33(4):143-61. doi: 10.3109/0167482X.2012.728649. PMID 23194018
- [Background] Dennis CL, Coghlan M, Vigod S. Can we identify mothers at-risk for postpartum anxiety in the immediate postpartum period using the State-Trait Anxiety Inventory? J Affect Disord. 2013 Sep 25;150(3):1217-20. doi: 10.1016/j.jad.2013.05.049. Epub 2013 Jun 10. PMID 23764383
- [Background] Kennedy SH, Lam RW, Cohen NL, Ravindran AV; CANMAT Depression Work Group. Clinical guidelines for the treatment of depressive disorders. IV. Medications and other biological treatments. Can J Psychiatry. 2001 Jun;46 Suppl 1:38S-58S. PMID 11441771
- [Background] World Health Organization. (WHO). Guidelines for Good Clinical Practice (GCP) for Trials on Pharmaceutical Products. WHO Technical Report Series, No. 850. (1995). 97-137
- [Background] Bricker, D & Squires, J. Ages and Stages Questionnaire. 3rd Ed. Baltimore, MD: Brookes Publishing; 2010.
- [Background] GlaxoSmithKline. GSK medicine: Bupropion and Paroxetine. Epidemiology study: Preliminary report on bupropion in pregnancy and the occurrence of cardiovascular and major congenital malformation (Study EPIP083). 2006; http://ctr.gsk.co.uk/summary/paroxetime/epip083.pdf.
- [Background] Vigod SN, Kurdyak PA, Dennis CL, Leszcz T, Taylor VH, Blumberger DM, Seitz DP. Transitional interventions to reduce early psychiatric readmissions in adults: systematic review. Br J Psychiatry. 2013 Mar;202(3):187-94. doi: 10.1192/bjp.bp.112.115030. PMID 23457182
- [Background] Demissie, K, Jospeh, KS, Dzakpasu, S. Perinatal Health Indicators for Canada: A Resource Manual. Public Health Agency of Canda, Canadian Perinatal Surveillance System. 2000; Ottawa, ON.
- [Background] Zuckerman B, Amaro H, Bauchner H, Cabral H. Depressive symptoms during pregnancy: relationship to poor health behaviors. Am J Obstet Gynecol. 1989 May;160(5 Pt 1):1107-11. doi: 10.1016/0002-9378(89)90170-1. PMID 2729387
- [Background] O'Hara MW, Swain AM. Rates and risk of postpartum depression: A meta-analysis. International Review of Psychiatry. 1996;8(1):37-54.
- [Derived] Vigod SN, Murphy KE, Dennis CL, Oberlander TF, Ray JG, Daskalakis ZJ, Blumberger DM. Transcranial direct current stimulation (tDCS) for depression in pregnancy: A pilot randomized controlled trial. Brain Stimul. 2019 Nov-Dec;12(6):1475-1483. doi: 10.1016/j.brs.2019.06.019. Epub 2019 Jun 19. PMID 31257092
- [Derived] Vigod S, Dennis CL, Daskalakis Z, Murphy K, Ray J, Oberlander T, Somerton S, Hussain-Shamsy N, Blumberger D. Transcranial direct current stimulation (tDCS) for treatment of major depression during pregnancy: study protocol for a pilot randomized controlled trial. Trials. 2014 Sep 18;15:366. doi: 10.1186/1745-6215-15-366. PMID 25234606